CLINICAL TRIAL: NCT04811248
Title: Respiratory Outcome of Infants With or Without Documented Wheezing During Bronchiolitis
Acronym: WheezOut
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200931; IDRCB: 2020-A01482-37 (Other: ANSM)
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-03

CONDITIONS: Wheezing; Asthma in Children
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: telephone call for parents of patients — telephone call for parents of patients aged 6 years old
  Other Names: one groupe of infants having a bronchiolitis

SUMMARY:
Hospital admission for infant bronchiolitis is associated with an increased risk of recurrent wheezing and subsequent asthma in childhood. In the literature, 17 to 60% of children will develop repeated wheezing (infant asthma in France). This highly variable incidence could be linked in part to the fact that the definition of bronchiolitis varies between continents. In Europe the usual definition is an acute and contagious viral infection which affects the bronchioles (small bronchi) of infants accompanied by coughing, rapid breathing and wheezing. In research studies, bronchiolitis must be associated with wheezing and / or crackles on auscultation in Europe, and wheezing imperatively in the USA. The diagnosis of wheezing is difficult, and medical agreement on auscultatory respiratory abnormalities is poor. We thus have developed a wheezing diagnostic tool using artificial intelligence processing of respiratory sound recordings by smartphone (Bokov P, Comput Biol Med 2016, DOI: 10.1016/j.compbiomed.2016.01.002). In a second larger bicentric study that included only infants suspected of bronchiolitis, our approach has consisted in obtaining a recording by smartphone but also by electronic stethoscope in order to allow deferred listening of the sounds (WheezSmart study). The objective of these studies was to obtain a formal diagnosis of wheezing, the current project aims to assess the benefit of this diagnosis. The main objective of this cross-sectional study is to determine whether the formal presence (diagnosis of wheezing from a recording of pulmonary auscultation) is associated with the risk of childhood asthma (diagnosis of asthma at 6 years) regardless of the usual risk factors (atopic / allergic terrain, exposure to smoking, recurrence of symptoms). The secondary objectives are to determine whether the formal presence of wheezing on auscultation is a risk factor for subsequent repeated wheezing (diagnosis of infant asthma) and for initial disease severity (bronchiolitis) compared to SpO2 and admission of the child to hospital. The interest in differentiating between high and low frequency sibilants will be evaluated also.

DETAILED DESCRIPTION:
Hospital admission for infant bronchiolitis is associated with an increased risk of recurrent wheezing and subsequent asthma in childhood. In the literature, 17 to 60% of children will develop repeated wheezing (infant asthma in France). This highly variable incidence could be linked in part to the fact that the definition of bronchiolitis varies between continents. In Europe the usual definition is an acute and contagious viral infection which affects the bronchioles (small bronchi) of infants accompanied by coughing, rapid breathing and wheezing. In research studies, bronchiolitis must be associated with wheezing and / or crackles on auscultation in Europe, and wheezing imperatively in the USA. The diagnosis of wheezing is difficult, and medical agreement on auscultatory respiratory abnormalities is poor. We thus have developed a wheezing diagnostic tool using artificial intelligence processing of respiratory sound recordings by smartphone (Bokov P, Comput Biol Med 2016, DOI: 10.1016/j.compbiomed.2016.01.002). In a second larger bicentric study that included only infants suspected of bronchiolitis, our approach has consisted in obtaining a recording by smartphone but also by electronic stethoscope in order to allow deferred listening of the sounds (WheezSmart study). The objective of these studies was to obtain a formal diagnosis of wheezing, the current project aims to assess the benefit of this diagnosis. The main objective of this cross-sectional study is to determine whether the formal presence (diagnosis of wheezing from a recording of pulmonary auscultation) is associated with the risk of childhood asthma (diagnosis of asthma at 6 years) regardless of the usual risk factors (atopic / allergic terrain, exposure to smoking, recurrence of symptoms). The secondary objectives are to determine whether the formal presence of wheezing on auscultation is a risk factor for subsequent repeated wheezing (diagnosis of infant asthma) and for initial disease severity (bronchiolitis) compared to SpO2 and admission of the child to hospital. The interest in differentiating between high and low frequency sibilants will be evaluated also. Population: Children from 3 to 7 years old. Inclusion criteria: • Children included in the WheezSmart study at Robert Debré Hospital • Diagnosis at inclusion of bronchiolitis • Telephone numbers of the 2 parents available • Informed parents who do not object to participation in research. Population of wheezsmart study: 281 children diagnosed with bronchiolitis at Robert Debré Hospital for whom we have a recording of respiratory sounds. Statistical analyses: Comparison of the proportions of infant asthma then asthma in the groups with and without wheezing (chi-square tests). For the two groups with and without wheezing, the SpO2 means and the hospital admission rate will be compared (t and chi-square test).

ELIGIBILITY:
Inclusion Criteria:

* Children included in the WheezSmart study at Robert Debré Hospital • Diagnosis at inclusion of bronchiolitis
* Telephone numbers of the 2 parents available
* Informed parents who do not object to participation in research.

Exclusion Criteria:

-

Ages: 3 Years to 7 Years | Sex: All
Age Groups: Child
Study Population: infant referred to emergency departement for bronchiolitis
Sampling Method: Non-Probability Sample
Enrollment: 281 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-01-08 (Estimated); Study Completion 2025-01-08 (Estimated)

PRIMARY OUTCOMES:
To assess whether diagnosis of wheezing from a recording of pulmonary auscultation is associated with the risk of childhood asthma | 1 year
  recording of asthma diagnosis and atopic, allergic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Plamen BOKOV, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided